CLINICAL TRIAL: NCT00450541
Title: The Experience of Fatigue for Patients With Cancer
Brief Title: Fatigue Experience in Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Other Study IDs: 2007-0004
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Fatigue; Interview; Questionnaire; Survey
MeSH Terms: conditions — Fatigue | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fatigue Questionnaire + Interview
  Interventions: Behavioral: Questionnaire; Behavioral: Interview

INTERVENTIONS:
Behavioral: Questionnaire — Four questionnaires taking 15-20 minutes total to complete.
  Other Names: Survey
Behavioral: Interview — Interview lasting about 30 minutes.

SUMMARY:
The goal of this research study is to learn what it is like when a patient with cancer has fatigue, as well as how these patients define fatigue. Researchers want to use this information to create questionnaires that may more accurately measure fatigue and its effects in patients with cancer.

DETAILED DESCRIPTION:
STUDY PARTICIPATION:

If you agree to take part in this study, you will be interviewed by a member of the study staff and then asked to complete a series of questionnaires and verbal (spoken) questions.

During the interview, you will be asked to describe what fatigue means to you and what it is like for you to have fatigue. The interview will take place while you are at M. D. Anderson receiving your routine care. You will be interviewed alone, and the information gathered during the interview will be kept strictly confidential. The interview will take about 30 minutes to complete. It will be audiotaped so that participants' responses can be fully analyzed.

You will then be asked to complete 4 questionnaires and answer 2 separate questions.

The first questionnaire will include questions about your personal identifying information (such as your age and marital status).

You will then be asked 1 question about your quality of life and another question about how well you are performing day-to-day activities.

You will then be asked to complete a second questionnaire in which you will rate your fatigue level and how fatigue interferes with your daily activities.

You will be asked to complete a third questionnaire about your opinion of the fatigue questionnaire (the second questionnaire). For example, you will be asked if the fatigue questionnaire was easy to understand and to complete. Learning your opinion about this questionnaire will help researchers learn what important questions may be missing from the questionnaire.

Finally, you will then be asked to complete a questionnaire that asks you to rate the severity of a list of 13 symptoms and how much these symptoms interfere with some of your daily activities.

The questionnaires and additional questions should take a total of 15-20 minutes to complete.

After you have completed the interview and questionnaires, a research assistant will review your electronic medical record to collect information about your disease and treatments.

LENGTH OF STUDY:

Your participation in this study will be over after you complete the interview, the questionnaires, and the additional questions.

This is an investigational study. Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Ability to speak and read English
3. Diagnosis of cancer, currently receiving treatment, receiving supportive care, or surviving after treatment
4. Self report of current experience of fatigue
5. Consent to participate
6. Patient from M. D. Anderson Cancer Center inpatient unit or outpatient clinic

Exclusion Criteria:

1. Inability to understand the intent of the study
2. Medical condition that would preclude participation in an interview session lasting 40 minutes
3. Diagnosis of active psychosis or severe cognitive impairment confirmed by the patient's attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer that may be experiencing fatigue.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2007-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Description of Cancer Patient Fatigue Experiences (Questionnaire + Interview Responses) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Loretta A. Williams, DSN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org